CLINICAL TRIAL: NCT07330973
Title: Effect of Transcutaneous Auricular Vagus Nerve Stimulation on Postoperative Pain in Patients Undergoing Complex Spinal Surgery: a Randomized Controlled Trial
Brief Title: Effects of taVNS on Postoperative Pain in Complex Spinal Surgery
Acronym: taVNS-cSSPain
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Principal Investigator, yu lina, Doctor, Second Affiliated Hospital, School of Medicine, Zhejiang University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2025-1950
Record Dates: First submitted 2025-12-17; First posted 2026-01-09 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2025-12

CONDITIONS: Postoperative Pain; Postoperative Pain in Orthopaedics; Postoperative Pain Management
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- taVNS group (Active Comparator): Paticipants in this arm will undergo a 60 minutes intervention of taVNS from one day before surgery to three days after surgery.
  Interventions: Device: transauricular auricular vagus nerve stimulation
- sham group (Sham Comparator): Paticipants in this arm will undergo a 60 minutes sham stimulation from one day before surgery to three days after surgery.
  Interventions: Device: transauricular auricular vagus nerve stimulation

INTERVENTIONS:
Device: transauricular auricular vagus nerve stimulation — Patients will receive five taVNS sessions, with each session lasting 60 minutes.
  Arms: taVNS group
Device: transauricular auricular vagus nerve stimulation — Patients will receive five sham taVNS sessions, with each session lasting 60 minutes.
  Arms: sham group

SUMMARY:
Transcutaneous auricular vagus nerve stimulation (taVNS) is a non-invasive, novel neuromodulation technique. Previous studies have demonstrated its safety and efficacy in chronic pain, mental disorders, and other diseases, but evidence regarding its use in acute postoperative pain remains limited. This project aims to explore the efficacy and safety of taVNS in managing acute pain after complex spinal surgery. This is a single-center, double-blind, randomized controlled clinical trial, planning to recruit 98 patients scheduled to undergo complex spinal surgery at the Second Affiliated Hospital of Zhejiang University School of Medicine. Participants will be randomly assigned to either the experimental group (taVNS stimulation) or the control group (sham stimulation). The experimental group will receive five stimulation sessions, each lasting one hour, from one day before surgery to three days after surgery. The primary outcome was opioid consumption within 72 hours postoperatively. Secondary outcomes included the maximum, minimum, and mean NRS on postoperative days 1, 2, and 3; NRS before and after each taVNS stimulation; time to first PCIA compression and number of PCA sessions within 3 days postoperatively; Hospital Anxiety and Depression Scale (HADS), Pittsburgh Sleep Quality Index (PSQI), and Quality of Recovery Scale (QoR15) on postoperative day 3; time to first flatus, and first bowel movement; and the incidence of chronic pain, HADS, PSQI, and QoR15 at 3 months postoperatively.

ELIGIBILITY:
Inclusion Criteria:

1. Patients undergoing elective general anesthesia for complex spinal surgeries
2. Age ≥ 18 years
3. ASA classification I-III

Exclusion Criteria:

1. Ulceration or infection of the auricle skin
2. Bradycardia (heart rate of < 60 beats/min） or third-degree atrioventricular block
3. Implanted cardiac pacemaker or other electronic devices
4. Mental disorders or long-term use of psychotropic medications
5. Severe hepatic and renal insufficiency
6. Unable to understand the content of the scale assessment or unable to cooperate with the scale assessment
7. Pregnant or lactating women
8. Expected reoperation during hospitalization
9. Expected to be transferred to the ICU after surgery
10. Participation in other concurrent clinical trials

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Estimated)
Dates: Start 2025-12-24 (Estimated); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Opioid consumption within 72 hours postoperatively | Within 72 hours postoperatively
  Researchers will record the dosage of opioids used by participants within 72 hours after surgery and convert it into morphine equivalents.

SECONDARY OUTCOMES:
Pain score | within 72 hours postoperatively
  Maximum, minimum, and mean NRS on postoperative days 1, 2, and 3, and NRS before and after taVNS stimulation.
Use of PCIA | Within 72 hours postoperatively
  Including the first compression time of PCA and times of PCA within 72 hours postoperatively
Hospital Anxiety and Depression Scale (HADS) within 3 months postoperatively | on the 3 months
  Assessed by HADS within 3 months postoperatively
Pittsburgh Sleep Quality Index (PSQI) within 3 months postoperatively | on the 3 months
  assessed by PSQI within 3 months postoperatively
Quality of Recovery Scale (QoR15) within 3 months postoperatively | on the 3 months
  Assessed by QoR15 within 3 months postoperatively
Incidence of chronic pain | at 3 months postoperatively
  Assessed by NRS at 3 months postoperatively
Functional recovery indicators | up to 2 weeks
  Including time to first flatus and time to first bowel movement
Length of hospital stay | up to 1 month
Adverse events | on the 3 months